CLINICAL TRIAL: NCT03293082
Title: The Effect of Continuous Glucose Monitoring Use on Glucose Variability in Preschool Children With Type 1 Diabetes
Brief Title: Preschool CGM Use and Glucose Variability in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: CGM-GV-Preschool- SI-01
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CGM ON — The period of time when continuous glucose monitoring was used, in edition to SMBG
Device: CGM OFF — The period of time when continuous glucose monitoring was not used, only SMBG

SUMMARY:
The objectives of this clinical study is to evaluate the efficacy continuous glucose monitoring (CGM) use on glucose variability (GV) in preschool children with T1D treated with CSII.

Downloads from CGM and CSII saved in pdf from will be retrospectively reviewed and analysed for all preschool children with type 1 diabetes in Slovenia. Glucose variability and other glycemic parameters will be analyzed separately for periods when CGM was used (CGM and SMBG data) and compared to periods when CGM was not used (SMBG only data).

ELIGIBILITY:
Inclusion Criteria:

1. Subject with Type 1 diabetes (> 6 months since diagnosis)
2. Insulin infusion pump CSII therapy for at least 3 months
3. Age ≤ 7 years
4. HbA1c at inclusion ≥ 6.5 and < 10
5. BMI SDS - below the 95th percentile for age

Exclusion Criteria:

1. Concomitant diseases that influence metabolic control
2. Participation in any other interventional study
3. Known or suspected allergy to trial products

Max Age: 7 Years | Sex: All
Age Groups: Child
Study Population: Population of preschool children with type 1 diabetes aged up to 7 years that were prescribed sensor use in the observational period.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Glucose variability | Three years
  Glucose variability as SD and CV of glucose levels measured with CGM and blood glucose

SECONDARY OUTCOMES:
Mean intersticial glucose | Three years
  Mean glucose as measured with CGM
Mean blood glucose | Three years
  Mean glucose as measured with SMBG
HbA1c | Three years
  glycosilated hemoglobin

CONTACTS AND LOCATIONS:
Locations (1):
- UMC - University Children's Hospital Ljubljana, Ljubljana, Slovenia